CLINICAL TRIAL: NCT04272515
Title: Molecular Characterization for Understanding Biliary Atresia
Acronym: CAVB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C19-36
Record Dates: First submitted 2020-01-28; First posted 2020-02-17 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: BA patients and their parents will be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BA patients and their parents (Experimental): * Collection of blood samples from BA patients and their parents
  * Collection of explanted liver tissue and skin biopsy of BA patients
  Interventions: Other: blood sampling; Other: skin biopsy sampling; Other: explanted liver of BA patients sampling

INTERVENTIONS:
Other: blood sampling — collection of blood sample for preparation of DNA
Other: skin biopsy sampling — preparation of primary cultures of dermal fibroblasts from skin biopsy sample
Other: explanted liver of BA patients sampling — cryoconservation of liver tissue for molecular analyses

SUMMARY:
Although considered a rare disease, Biliary Atresia (BA) is the leading cause of neonatal cholestasis and liver transplantation in children. Little is known about the molecular mechanisms that drive BA. The purpose of this study is to collect the fluid samples, explanted liver tissue samples and dermal biopsy samples to enable investigators to perform the genetic and molecular analyses that might point to the gene(s) and cellular pathway involved in etiology of BA disease.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a disease characterized by intra- and extra-hepatic bile duct obstruction diagnosed in the neonatal period. If left untreated, this obstruction leads to biliary cirrhosis and early death. Although considered a rare disease (between 1/15,000 and 1/20000 births), it is the leading cause of neonatal cholestasis and liver transplantation in children. The reasons for this obstruction are still poorly known and might involve several factors (immune, infectious and possible toxin effect). The accumulating evidence point to genetic factors involved, yet they are not of the classic monogenic or Mendelian types. The purpose of this study is to collect the fluid samples, explanted liver tissue samples and dermal biopsy samples to enable investigators to perform the genetic and molecular analyses that might point to the gene(s) and cellular pathway involved in etiology of BA disease.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of biliary atresia in patients
* parents of BA patients

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-07 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2032-02-07 (Estimated)

PRIMARY OUTCOMES:
To identify the molecular mechanisms implicated in the etiology of BA | 10 Years
  To identify gene(s) and cellular pathways affected in cells and liver tissue of BA patients: sequencing experiments

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Necker enfants malades, Paris, De
  - PRC Inserm, Paris

IPD SHARING:
Plan to Share IPD: No